CLINICAL TRIAL: NCT00720733
Title: A Positive Affect Intervention for Those Recently Diagnosed With HIV
Brief Title: Intervention for (Those) Recently Informed of Seropositive Status (IRISS)
Acronym: IRISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RMH084723A; 1RO1MHO84723-01
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: HIV; Mood; Emotion; Coping; Aids; Affect; Adults; Diagnosed
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Skills Building Group
  Interventions: Behavioral: Skills-Building Intervention
- 2 (Active Comparator): Personal Interview Group
  Interventions: Behavioral: Personal Interview Group

INTERVENTIONS:
Behavioral: Skills-Building Intervention — A 5-week intervention including 5 weekly sessions covering 8 varied coping skills with daily home practice. The skills are: 1) noting daily positive events; 2) capitalizing on positive events; 3) gratitude; 4) mindfulness; 5) positive reappraisal; 6) focusing on personal strengths; 7) setting and working toward attainable goals; and 8) small acts of kindness. Sessions are 1 hour long and include approximately 30 minutes per day.
  Arms: 1
Behavioral: Personal Interview Group — There are 5 weekly sessions which will be approximately one hour long and will consist of personal interview. The interviews will include both quantitative and qualitative questions. Each session will have a separate theme including: Life 1) History; 2) Health History; 3) Personality; 4) Social Networking; and, 5) Meaning & Purpose.
  Arms: 2

SUMMARY:
An intervention designed to increase positive affect in a population newly diagnosed with HIV will be effective at improving affect and HIV-related outcomes such as mental and physical health, coping and coping resources.

DETAILED DESCRIPTION:
The study is a randomized controlled trial of a 5-session positive affect skills intervention compared to an attention-matched control condition. Participants will be 200 men and women who have tested positive for HIV within the past 12 weeks. Both intervention and control sessions will be approximately one hour long and will be administered one-on-one by trained facilitators. Both groups will have daily home practice over the 5 weeks of the intervention. At the end of the assessment period, participants in the control condition will have the opportunity to attend a ½ day group session that provides a condensed version of the positive affect skills taught in the intervention condition. Participants will complete assessments at four points and CD4 and viral load assays will be run at 3 time points.

ELIGIBILITY:
Inclusion Criteria:

* have been informed they were HIV positive within the past 12 weeks
* speak English or Spanish
* be 18 years or older
* have the ability to provide informed consent to be a research participant.

Exclusion Criteria:

* inability to provide informed consent, as evidenced by cognitive impairment as assessed by trained interviewers and confirmed by a licensed clinical psychologist
* active psychosis as assessed by trained interviewers and confirmed by clinical psychologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of the Intervention for those Recently Informed of their Seropositive Status (IRISS) for increasing the frequency and intensity of positive affect in men and women newly diagnosed with HIV. | During the intervention and at 5- 10- and 15-months after diagnosis.

SECONDARY OUTCOMES:
Effects on outcomes and if increases in positive affect are responsible for improvements; effects of individual facets on affect and outcomes; and, evaluate extent to which personality, se status, race/ethn, & stress level, moderate effects on outcomes. | At 15 months post diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Judith T Moskowitz, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Moskowitz JT, Carrico AW, Duncan LG, Cohn MA, Cheung EO, Batchelder A, Martinez L, Segawa E, Acree M, Folkman S. Randomized controlled trial of a positive affect intervention for people newly diagnosed with HIV. J Consult Clin Psychol. 2017 May;85(5):409-423. doi: 10.1037/ccp0000188. Epub 2017 Mar 23. PMID 28333512